CLINICAL TRIAL: NCT01574703
Title: A Phase 4, Non-treatment Follow-up For Cardiac Assessments Following Use Of Smoking Cessation Treatments In Subjects With And Without A History Of Psychiatric Disorders
Brief Title: Study To Evaluate Cardiac Assessments Following Different Treatments Of Smoking Cessation Medications In Subjects With And Without Psychiatric Disorders.
Acronym: CATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: A3051148; 2011-005513-37 (EudraCT Number); CATS (Other: Alias Study Number)
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; psychiatric disease; cardiovascular events
MeSH Terms: conditions — Smoking Cessation; Mental Disorders | interventions — Varenicline; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo (Experimental)
  Interventions: Drug: placebo
- varenicline (Experimental)
  Interventions: Drug: varenicline tartrate
- bupropion (Experimental)
  Interventions: Drug: bupropion hydrochloride
- Nicotine Replacement Therapy Patch (Experimental)
  Interventions: Drug: Nicotine Replacement Therapy Patch

INTERVENTIONS:
Drug: placebo — All dosing to have taken place per study A3051123
  Arms: placebo
Drug: varenicline tartrate — All dosing to have taken place per study A3051123
  Other Names: Chantix; Champix
  Arms: varenicline
Drug: bupropion hydrochloride — All dosing to have taken place per study A3051123
  Other Names: Zyban
  Arms: bupropion
Drug: Nicotine Replacement Therapy Patch — All dosing to have taken place per study A3051123
  Other Names: NRT
  Arms: Nicotine Replacement Therapy Patch

SUMMARY:
Non-treatment extension to study A3051123, aimed at collecting data on cardiovascular safety for all participants in the A3051123 trial for an additional 28 weeks, allowing for a total of 52 weeks of cardiovascular safety data collection.

DETAILED DESCRIPTION:
This study is an extension protocol for study A3051123. No treatment is provided during this study. This study is to monitor for cardiovascular events 28 weeks after completion of A3051123. This study is an extension protocol for study A3051123. No treatment is provided during this study. This study is to monitor for cardiovascular events 28 weeks after completion of A3051123.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if they were randomized to study A3051123.

Exclusion Criteria:

* Participation in study A3051123 ceased (ie, withdrew consent, lost to follow-up, etc) prior to final visit of study A3051123.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4595 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (133):
- United States (64):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Pharmacology Research Institute, Encino, California
  - Synergy Clinical Research Center of Escondido, Escondido, California
  - Sun Valley Research Center, Imperial, California
  - Omega Clinical Trials, La Habra, California
  - Pacific Treatment and Research Center, La Jolla, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute (PRI), Newport Beach, California
  - North County Clinical Research, Oceanside, California
  - NRC Research Institute, Orange, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - University of Colorado Anschutz Medical Campus Behavioral Health and Wellness Program, Aurora, Colorado
  - Western Affiliated Research Institute, Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Broward Research Group, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - Ocala Psychiatric Associates, Ocala, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Baber Research Group Incorporated, Naperville, Illinois
  - Davis Clinic, Incorporated, Indianapolis, Indiana
  - American Health Network of IN, LLC, Indianapolis, Indiana
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Incorporated, Lexington, Kentucky
  - Kentucky Research Group, Louisville, Kentucky
  - The Center for Sexual Health, Metairie, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Milford Emergency Associates, Incorporated, Milford, Massachusetts
  - University of Minnesota - TC, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - CRI Worldwide, LLC, Marlton, New Jersey
  - Global Medicinal Institutes, LLC; Princeton Medical Institute, Princeton, New Jersey
  - SPRI Clinical Trails LLC, Brooklyn, New York
  - Regional Clinical Research, Incorporated, Endwell, New York
  - PMG Research of Raleigh, LLC, Cary, North Carolina
  - Wake Internal Medicine Consultants, Inc, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Southeastern PA Medical Institute, Broomall, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - Lincoln Research, LLC, Lincoln, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Clinical Neuroscience Solutions,Inc, Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - James G. Kyser, MD, Nashville, Tennessee
  - Future Search Clinical Trials, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Clinical Research Associates of Tidewater, Inc, Norfolk, Virginia
- Argentina (2):
  - Centro de Investigacion Clinica WM, Capital Federal, Buenos Aires
  - Centro Medico Dra. De Salvo, Buenos Aires, Buenos Aires F.D.
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia
- Brazil (3):
  - Hospital Sao Lucas da PUCRS - Uniao Brasileira de Educacao e Assistencia, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - Pontifícia Universidade Católica de Campinas - Campus II, Campinas, São Paulo
  - Jaqueline Scholz Issa e Mario Issa de cardiologia Ltda, São Paulo, São Paulo
- Bulgaria (10):
  - Mental Health Center "Prof. Dr. Ivan Temkov-Bourgas" Ltd., Burgas, Bourgas
  - MHAT "Dr. Hristo Stambolski" Ltd., Kazanlak
  - NPH "Sv. Ivan Rilski", Novi Iskar
  - UMHAT "Dr. Georgi Stranski" Ltd., Pleven
  - UMHAT "Sveti Georgi" Ltd., Plovdiv
  - SHATPPD - Ruse Ltd., Rousse
  - Mental Health Center - Ruse Ltd., Rousse
  - MHATNP "Sveti Naum" Ltd., Sofia
  - MHATNP Sveti Naum SJsc., Sofia
  - SHATPD - Troyan Ltd., Troyan Municipality
- Canada (6):
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Medical Research Associates, Mississauga, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Chile (2):
  - Hospital Regional de Talca, Unidad de Enfermedades Respiratorias, Talca, Maule Region
  - Centro Respiratorio Integral (CENRESIN Ltda.), Quillota, Valparaiso, V Region
- Denmark (2):
  - CCBR A/S, Ballerup Municipality
  - CCBR A/S, Vejle
- Finland (6):
  - Mehiläinen Leppävaara, Espoo, Finland
  - Savon Psykiatripalvelu Oy, Kuopio, Finland
  - Oulu Mentalcare Oy, Oulu, Finland
  - Mehiläinen Nummela, Nummela
  - Porin Lääkäritalo Oy, Pori
  - PEL, Psykiatrian ErikoisLääkärit, Turku
- Germany (7):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Ludwig Maximilians-Universitaet Muenchen, Munich, Bavaria
  - Klinische Forschung Hamburg GmbH, Hamburg, Hamburg
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - emovis GmbH, Berlin
  - ZSL - Zentrum fuer Medizinische Studien Leipzig GmbH, Leipzig
  - Universitaetsklinik Tuebingen, Klinik fuer Psychiatrie und Psychotherapie, Tübingen
- Mexico (2):
  - Consultorios de Medicina Especializada del Sector Privado, México, Mexico Df
  - Centro de Estudios Clinicos y Especialidades Medicas S.C., Monterrey, Nuevo León
- Lakeland Clinical Trials, Rotorua, New Zealand
- Russia (7):
  - FSBI "Federal Medical Research Center of Psychiatry and Addiction Medicine", Moscow
  - Moscow State Public Healthcare Institution Mental Clinical Hospital #1 n.a. N.A. Alexeeva, Moscow
  - Clinical Mental Hospital #12 of Moscow Healthcare Department, Moscow
  - Clinical Psychiatric Hospital #1 of Nizhni Novgorod, Nizhny Novgorod
  - St. Petersburg State Healthcare Institution, St. Nikolay Chudotvorets Mental Hospital, Saint Petersburg
  - FSBI "Saint-Petersburg Scientific Research Psychoneurological Institute n.a. V.M. Bekhterev", Saint Petersburg
  - State Healthcare Institution of St.Petersburg "Psychoneurological Dispensary #2, Saint Petersburg
- Slovakia (5):
  - Psychiatricka ambulancia, Mentum, s.r.o., Bratislava
  - Nestatna psychiatricka ambulancia, MUDr. Livia Vavrusova, PhD, Bratislava
  - Psychiatricka ambulancia MUDr. Nada Kuriackova, s.r.o., Levice
  - Psychiatricka ambulancia, PsychoLine s.r.o., Rimavská Sobota
  - Nemocnica s poliklinikou sv. Barbory Roznava a.s., Rožňava
- South Africa (9):
  - Flexivest Fourteen Research Center, Bellville, Cape Town
  - Worthwhile Clinical Trials, Benoni, Johannesburg, Gauteng
  - Soweto Clinical Trials Centre, Johannesburg, Gauteng
  - Midrand Medical Centre, Midrand, Gauteng
  - I Engelbrecht Research Pty. Ltd, Pretoria, Gauteng
  - Vista Clinic, Pretoria, Gauteng
  - Private Practice, Durban, Kwa-zulu Natal, South Africa
  - Randles Road Medical Centre, Durban, KwaZulu-Natal
  - Dr John O'Brien Incorporated, Cape Town, Western Cape
- Spain (6):
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital General Universitari Vall D'Hebron, Barcelona, Barcelona
  - Hospital Clinic I Provincial, Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres, Caceres
  - Unidad Especializada En Tabaquismo de La Comunidad de Madrid, Madrid, Madrid
  - Centro de Salud Torrero-La Paz., Zaragoza, Zaragoza

REFERENCES:
- [Derived] Benowitz NL, Pipe A, West R, Hays JT, Tonstad S, McRae T, Lawrence D, St Aubin L, Anthenelli RM. Cardiovascular Safety of Varenicline, Bupropion, and Nicotine Patch in Smokers: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):622-631. doi: 10.1001/jamainternmed.2018.0397. PMID 29630702
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051148&StudyName=Study%20To%20Evaluate%20Cardiac%20Assessments%20Following%20Different%20Treatments%20Of%20Smoking%20Cessation%20Medications%20In%20Subjects%20With%20And%20without%20Psychiatr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 6293 participants who completed the parent study NCT01456936 as per protocol, a total of 4595 participants enrolled into this study NCT01574703 from 132 centers in 16 countries.
Pre-assignment Details: This is a non-treatment extension study of parent study NCT01456936. No study drug was provided in this extension phase. However, cardiovascular events that occurred during parent study NCT01456936 when participants received varenicline(N=2016), bupropion(N=2006),NRT(N=2022), or placebo(N=2014) in a triple-dummy design were analyzed in this study.
Groups:
- Varenicline: This was the non-treatment extension study of parent study NCT01456936. No study drug was provided during this extension phase. However, Cardiovascular events that occurred during parent study NCT01456936 when participants received varenicline in a triple-dummy design were analyzed as part of this study.
- Bupropion: This was the non-treatment extension study of parent study NCT01456936. No study drug was provided during this extension phase. However, Cardiovascular events that occurred during parent study NCT01456936 when participants received bupropion in a triple-dummy design were analyzed as part of this study.
- Nicotine Replacement Therapy (NRT) Patch: This was the non-treatment extension study of parent study NCT01456936. No study drug was provided during this extension phase. However, Cardiovascular events that occurred during parent study NCT01456936 when participants received NRT patch in a triple-dummy design were analyzed as part of this study.
- Placebo: This was the non-treatment extension study of parent study NCT01456936. No study drug was provided during this extension phase. However, Cardiovascular events that occurred during parent study NCT01456936 when participants received placebo in a triple-dummy design were analyzed as part of this study.
Period: Overall Study
Arm/Group | Varenicline | Bupropion | Nicotine Replacement Therapy (NRT) Patch | Placebo
Started | 1192 | 1166 | 1116 | 1121
Completed | 1067 | 1054 | 1011 | 1007
Not Completed | 125 | 112 | 105 | 114
Not completed — Adverse Event | 0 | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Unspecified Reason | 27 | 15 | 20 | 16
Not completed — Withdrawal by Subject | 53 | 52 | 36 | 61
Not completed — Met Withdrawal Criteria | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 43 | 41 | 46 | 35
Not completed — Death | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The term Baseline visit refers to the Baseline (Week 0) visit of the parent study NCT01456936. The safety population included all participants who received at least one dose of study drug in NCT01456936 parent study. The below Baseline characteristics (age, gender) are presented for all participants who entered study NCT01574703.
Groups:
- NRT Patch: This was the non-treatment extension study of parent study NCT01456936. No study drug was provided during this extension phase. However, Cardiovascular events that occurred during parent study NCT01456936 when participants received NRT patch in a triple-dummy design were analyzed as part of this study.
- Total: Total of all reporting groups
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo | Total
Number analyzed (Participants) | 1192 | 1166 | 1116 | 1121 | 4595
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (12.2) | 47.7 (12.5) | 48.3 (11.9) | 47.5 (12.2) | 47.9 (12.2)
Gender [Count of Participants; unit: Participants]
  Female | 659 | 648 | 623 | 621 | 2551
  Male | 533 | 518 | 493 | 500 | 2044

OUTCOME MEASURES:

1. Primary Outcome: Time to Occurrence of Major Adverse Cardiovascular Event (MACE) During Treatment Period (up to Date of Last Dose of Study Drug) in Study NCT01456936.
Description: This is an adjudicated endpoint. MACE is defined as a cardiovascular death, a non-fatal myocardial infarction or a non-fatal stroke evaluated during the treatment phase (up to date of last dose of study drug). The measure type mentioned in the outcome data table is Hazard Ratio relative to Placebo.
Time Frame: Baseline to last dose of study drug in parent study NCT01456936 (up to 12 weeks).
Population: The safety analysis set is defined as all participants that received at least one partial dose of study drug during the parent study NCT01456936.
Measure: Number (95% Confidence Interval); unit: Unitless
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
Unitless | 0.29 [0.05 to 1.68] | 0.50 [0.10 to 2.50] | 0.29 [0.05 to 1.70] | NA [NA to NA] — Hazard ratio relative to Placebo.
Statistical Analysis 1: Comparison: Varenicline vs Bupropion vs NRT Patch vs Placebo; Statistical analysis for overall treatment comparison; Test type: Superiority or Other; p = 0.37, Log Rank — P-value for the treatment effect from the Log-Rank test stratified by Cohort

2. Secondary Outcome: Time to MACE up to Date of Last Dose of Study Drug Plus 30 Days Follow-up in Study NCT01456936.
Description: This is an adjudicated endpoint. MACE is defined as a cardiovascular death, a non-fatal myocardial infarction or a non-fatal stroke evaluated during the treatment phase (up to date of last dose of study drug) plus 30 days follow-up. The measure type mentioned in the outcome data table is Hazard Ratio.
Time Frame: Baseline to last dose of study drug in parent study NCT01456936 (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Unitless
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
Unitless | 0.29 [0.05 to 1.70] | 0.51 [0.10 to 2.51] | 0.50 [0.10 to 2.48] | NA [NA to NA] — Hazard ratio relative to Placebo.
Statistical Analysis 1: Comparison: Varenicline vs Bupropion vs NRT Patch vs Placebo; Statistical analysis for overall treatment comparison; Test type: Superiority or Other; p = 0.53, Log Rank — P-value for the treatment effect from the Log-Rank test stratified by Cohort

3. Secondary Outcome: Time to MACE Until the End of Study NCT01574703.
Description: This is an adjudicated endpoint. MACE is defined as a cardiovascular death, a non-fatal myocardial infarction or a non-fatal stroke evaluated until end of study. The measure type mentioned in the outcome data table is Hazard Ratio.
Time Frame: Baseline until end of study (end of study is defined as last visit in study NCT01574703 [up to Week 52], or in study NCT01456936 [up to 24 Weeks] for those participants not enrolled into study NCT01574703).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Unitless
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
Unitless | 0.39 [0.12 to 1.27] | 1.09 [0.42 to 2.83] | 0.75 [0.26 to 2.13] | NA [NA to NA] — Hazard ratio relative to Placebo.
Statistical Analysis 1: Comparison: Varenicline vs Bupropion vs NRT Patch vs Placebo; Statistical analysis for overall treatment comparison; Test type: Superiority or Other; p = 0.34, Log Rank — P-value for the treatment effect from the Log-Rank test stratified by Cohort

4. Secondary Outcome: Incidence of MACE Assessed During Treatment Period (up to Date of Last Dose of Study Drug) in Study NCT01456936.
Description: This is an adjudicated endpoint. MACE is defined as a cardiovascular death, a non-fatal myocardial infarction or a non-fatal stroke evaluated during the treatment phase (up to date of last dose of study drug).
Time Frame: Baseline to last dose of study drug in parent study NCT01456936 (up to 12 weeks).
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants | 0.05 | 0.10 | 0.05 | 0.20
Statistical Analysis 1: Comparison: Varenicline vs Bupropion; Statistical analysis between Varenicline and Bupropion; Test type: Superiority or Other; p = 0.8375, Regression, Logistic — P-values are for the risk differences of pairwise comparisons based on the logistic regression model with terms Baseline Cardiovascular Risk, treatment, cohort, region, and treatment by cohort interaction; Risk Difference (RD) = -0.49, 95% CI 2-sided [-5.22 to 4.23]
Statistical Analysis 2: Comparison: Varenicline vs NRT Patch; Statistical analysis between Varenicline and NRT patch; Test type: Superiority or Other; p = 0.9780, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.07, 95% CI 2-sided [-5.20 to 5.05]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis between Varenicline and Placebo; Test type: Superiority or Other; p = 0.6142, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -1.13, 95% CI 2-sided [-5.54 to 3.27]
Statistical Analysis 4: Comparison: Bupropion vs NRT Patch; Statistical analysis between Bupropion and NRT patch; Test type: Superiority or Other; p = 0.8602, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.42, 95% CI 2-sided [-4.28 to 5.13]
Statistical Analysis 5: Comparison: Bupropion vs Placebo; Statistical analysis between Bupropion and Placebo; Test type: Superiority or Other; p = 0.7217, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.64, 95% CI 2-sided [-4.15 to 2.88]
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Statistical analysis between NRT patch and Placebo; Test type: Superiority or Other; p = 0.6322, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -1.06, 95% CI 2-sided [-5.41 to 3.28]

5. Secondary Outcome: Incidence of MACE + Assessed During Treatment Period (up to Date of Last Dose of Study Drug) in Study NCT01456936.
Description: This is an adjudicated endpoint. MACE + is defined as any MACE or a new onset or worsening peripheral vascular disease (PVD) requiring intervention, a need for coronary revascularization, or hospitalization for unstable angina.
Time Frame: Baseline to last dose of study drug in parent study NCT01456936 (up to 12 weeks).
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants | 0.25 | 0.20 | 0.10 | 0.25
Statistical Analysis 1: Comparison: Varenicline vs Bupropion; Statistical analysis between Varenicline and Bupropion; Test type: Superiority or Other; p = 0.9687, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.07, 95% CI 2-sided [-3.48 to 3.34]
Statistical Analysis 2: Comparison: Varenicline vs NRT Patch; Statistical analysis between Varenicline and NRT patch; Test type: Superiority or Other; p = 0.7905, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.56, 95% CI 2-sided [-3.58 to 4.70]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis between Varenicline and Placebo; Test type: Superiority or Other; p = 0.8962, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.21, 95% CI 2-sided [-3.36 to 2.94]
Statistical Analysis 4: Comparison: Bupropion vs NRT Patch; Statistical analysis between Bupropion and NRT patch; Test type: Superiority or Other; p = 0.7767, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.63, 95% CI 2-sided [-3.72 to 4.98]
Statistical Analysis 5: Comparison: Bupropion vs Placebo; Statistical analysis between Bupropion and Placebo; Test type: Superiority or Other; p = 0.9260, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.14, 95% CI 2-sided [-3.13 to 2.85]
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Statistical analysis between NRT patch and Placebo; Test type: Superiority or Other; p = 0.7113, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.77, 95% CI 2-sided [-4.85 to 3.31]

6. Secondary Outcome: Incidence of MACE Assessed up to Date of Last Dose of Study Drug Plus 30 Days Follow-up in Study NCT01456936.
Description: This is an adjudicated endpoint. MACE is defined as a cardiovascular death, a non-fatal myocardial infarction or a non-fatal stroke evaluated during the treatment phase (up to date of last dose of study drug) plus 30 days follow-up.
Time Frame: Baseline to last dose of study drug in parent study NCT01456936 (up to 12 weeks) plus 30 days follow-up.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants | 0.05 | 0.10 | 0.10 | 0.20
Statistical Analysis 1: Comparison: Varenicline vs Bupropion; Statistical analysis between Varenicline and Bupropion; Test type: Superiority or Other; p = 0.8117, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.57, 95% CI 2-sided [-5.27 to 4.13]
Statistical Analysis 2: Comparison: Varenicline vs NRT Patch; Statistical analysis between Varenicline and NRT patch; Test type: Superiority or Other; p = 0.7303, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.78, 95% CI 2-sided [-5.21 to 3.65]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis between Varenicline and Placebo; Test type: Superiority or Other; p = 0.5946, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -1.20, 95% CI 2-sided [-5.60 to 3.21]
Statistical Analysis 4: Comparison: Bupropion vs NRT Patch; Statistical analysis between Bupropion and NRT patch; Test type: Superiority or Other; p = 0.9200, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.21, 95% CI 2-sided [-4.27 to 3.85]
Statistical Analysis 5: Comparison: Bupropion vs Placebo; Statistical analysis between Bupropion and Placebo; Test type: Superiority or Other; p = 0.7236, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.62, 95% CI 2-sided [-4.09 to 2.84]
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Statistical analysis between NRT patch and Placebo; Test type: Superiority or Other; p = 0.8201, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.42, 95% CI 2-sided [-4.01 to 3.17]

7. Secondary Outcome: Incidence of MACE+ Assessed up to Date of Last Dose of Study Drug Plus 30 Days Follow-up in Study NCT01456936.
Description: This is an adjudicated endpoint. MACE + is defined as any MACE or a new onset or worsening PVD requiring intervention, a need for coronary revascularization, or hospitalization for unstable angina.
Time Frame: Baseline to last dose of study drug in parent study NCT01456936 (up to 12 weeks) plus 30 days follow-up.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants | 0.25 | 0.20 | 0.15 | 0.35
Statistical Analysis 1: Comparison: Varenicline vs Bupropion; Statistical analysis between Varenicline and Bupropion; Test type: Superiority or Other; p = 0.8932, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.21, 95% CI 2-sided [-3.22 to 2.81]
Statistical Analysis 2: Comparison: Varenicline vs NRT Patch; Statistical analysis between Varenicline and NRT patch; Test type: Superiority or Other; p = 0.8747, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.23, 95% CI 2-sided [-3.09 to 2.63]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis between Varenicline and Placebo; Test type: Superiority or Other; p = 0.6710, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.60, 95% CI 2-sided [-3.35 to 2.15]
Statistical Analysis 4: Comparison: Bupropion vs NRT Patch; Statistical analysis between Bupropion and NRT patch; Test type: Superiority or Other; p = 0.9886, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.02, 95% CI 2-sided [-3.32 to 3.27]
Statistical Analysis 5: Comparison: Bupropion vs Placebo; Statistical analysis between Bupropion and Placebo; Test type: Superiority or Other; p = 0.7631, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.39, 95% CI 2-sided [-2.92 to 2.14]
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Statistical analysis between NRT patch and Placebo; Test type: Superiority or Other; p = 0.8022, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.37, 95% CI 2-sided [-3.23 to 2.50]

8. Secondary Outcome: Incidence of MACE Assessed Until End of Study NCT01574703.
Description: This is an adjudicated endpoint. MACE is defined as a cardiovascular death, a non-fatal myocardial infarction or a non-fatal stroke evaluated until end of study.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants | 0.15 | 0.45 | 0.30 | 0.40
Statistical Analysis 1: Comparison: Varenicline vs Bupropion; Statistical analysis between Varenicline and Bupropion; Test type: Superiority or Other; p = 0.6441, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.91, 95% CI 2-sided [-4.78 to 2.96]
Statistical Analysis 2: Comparison: Varenicline vs NRT Patch; Statistical analysis between Varenicline and NRT patch; Test type: Superiority or Other; p = 0.7327, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.69, 95% CI 2-sided [-4.63 to 3.26]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis between Varenicline and Placebo; Test type: Superiority or Other; p = 0.6109, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.99, 95% CI 2-sided [-4.80 to 2.82]
Statistical Analysis 4: Comparison: Bupropion vs NRT Patch; Statistical analysis between Bupropion and NRT patch; Test type: Superiority or Other; p = 0.8707, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.22, 95% CI 2-sided [-2.48 to 2.93]
Statistical Analysis 5: Comparison: Bupropion vs Placebo; Statistical analysis between Bupropion and Placebo; Test type: Superiority or Other; p = 0.9531, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.08, 95% CI 2-sided [-2.63 to 2.48]
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Statistical analysis between NRT patch and Placebo; Test type: Superiority or Other; p = 0.8262, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.30, 95% CI 2-sided [-2.99 to 2.39]

9. Secondary Outcome: Incidence of MACE+ Assessed Until End of Study NCT01574703.
Description: This is an adjudicated endpoint. MACE+ is defined as any MACE or a new onset or worsening PVD requiring intervention, a need for coronary revascularization, or hospitalization for unstable angina.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants | 0.50 | 0.75 | 0.49 | 0.60
Statistical Analysis 1: Comparison: Varenicline vs Bupropion; Statistical analysis between Varenicline and Bupropion; Test type: Superiority or Other; p = 0.6105, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.59, 95% CI 2-sided [-2.84 to 1.67]
Statistical Analysis 2: Comparison: Varenicline vs NRT Patch; Statistical analysis between Varenicline and NRT patch; Test type: Superiority or Other; p = 0.7895, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.32, 95% CI 2-sided [-2.65 to 2.01]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis between Varenicline and Placebo; Test type: Superiority or Other; p = 0.6804, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.48, 95% CI 2-sided [-2.75 to 1.80]
Statistical Analysis 4: Comparison: Bupropion vs NRT Patch; Statistical analysis between Bupropion and NRT patch; Test type: Superiority or Other; p = 0.8127, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.27, 95% CI 2-sided [-1.95 to 2.49]
Statistical Analysis 5: Comparison: Bupropion vs Placebo; Statistical analysis between Bupropion and Placebo; Test type: Superiority or Other; p = 0.9218, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.11, 95% CI 2-sided [-2.04 to 2.25]
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Statistical analysis between NRT patch and Placebo; Test type: Superiority or Other; p = 0.8841, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.16, 95% CI 2-sided [-2.32 to 2.00]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Week 24 visit of study NCT01456936 until the end of study (i.e. Week 52 or date of discontinuation, as applicable).
Description: Safety analysis set: Participants that received at least one dose of study drug during the parent study (i.e., NCT01456936). Four deaths (completed suicide, death, myocardial infarction and upper gastrointestinal haemorrhage) are listed as serious AEs below, included events that began 31 days after the last dose of study drug in study NCT01456936.
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Serious Adverse Events (participants affected / at risk) | 34/1192 | 39/1166 | 43/1116 | 41/1121
Other Adverse Events (participants affected / at risk) | 165/1192 | 160/1166 | 116/1116 | 143/1121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=1192) | Bupropion (N=1166) | NRT Patch (N=1116) | Placebo (N=1121)
Acute myocardial infarction (Cardiac disorders) | 0 | 4 | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 2
Coronary artery disease (Cardiac disorders) | 2 | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 1 | 0 | 0
Endocrine ophthalmopathy (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Haemorrhagic fever with renal syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 0
Post procedural infection (Infections and infestations) | 1 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatosplenic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Morton's neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 1 | 2
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 1 | 0
Major depression (Psychiatric disorders) | 2 | 1 | 0 | 2
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 2 | 1 | 2
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Drug detoxification (Surgical and medical procedures) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=1192) | Bupropion (N=1166) | NRT Patch (N=1116) | Placebo (N=1121)
Nasopharyngitis (Infections and infestations) | 103 | 78 | 69 | 81
Upper respiratory tract infection (Infections and infestations) | 63 | 84 | 48 | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.